CLINICAL TRIAL: NCT00533078
Title: Lipid Use, Nutrition, and Colitis in Patients With Hematological Malignancies (LUNCH1)
Brief Title: Lipid Use, Nutrition, and Colitis in Patients With Hematological Malignancies
Acronym: LUNCH1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Johannes Buekki, MD, University Hospital Inselspital, Berne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007DR2232; 1345 (institution); 120/07 (ethics review board)
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Colitis; Mucositis; AML
Keywords: omega3 fatty acid; parenteral nutrition; chemotherapy; infection; neutropenia
MeSH Terms: conditions — Colitis; Mucositis; Hyperphagia; Infections; Neutropenia | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Dietary Supplement: omegaven

INTERVENTIONS:
Dietary Supplement: omegaven — Trial participants are prescribed TPN by the attending physician as soon as indicated, which will be administered via a central venous line over a time period of approximately 20 hours per day. The formulation given to all patients is Nutriflex lipid spezial®, an emulsion containing the full supply of carbohydrates, amino acids and lipids (SO:MCT = 1:1) with a total energy content of 2215 kcal in a 1875 ml volume, see Investigator's Brochure. In addition, they receive daily infusional Omegaven® 100 ml over 4 hours, which equal FO 10 g/d or omega-3 PUFA 3-6 g/d.

SUMMARY:
In patients with acute myelogenous leukemia (AML), a high proportion will suffer from inflammation of the large bowel (colitis) during their intensive treatment. As there is no standard treatment available for this potentially lifethreatening condition, the investigators focus on the role of parenteral nutrition which these patients inevitably require. Preclinical and clinical data have shown strong anti-inflammatory properties of fish oil preparations containing poly-unsaturated omega3 fatty acids (PUFA) as opposed to other lipid fractions. There may be a therapeutic benefit of adding omega3 PUFA to standard nutrition in patients with chemotherapy-induced colitis. In this small phase II study, the investigators address the effectiveness of this approach to reduce the incidence and severity of colitis in AML patients.

DETAILED DESCRIPTION:
Experimental and clinical data attribute multiple anti-inflammatory effects to a diet enriched in omega-3 PUFA containing oils, mainly FO. These effects are mediated by their active metabolites, the EPA- and DHA-derived eicosanoids, which antagonize the predominantly pro-inflammatory derivates of omega-6 PUFA origin. In cardiovascular disease these data are supported by several large-scale trials, but there also is growing evidence of beneficial effects of an omega-3 PUFA rich diet in GI conditions such as postoperative trauma and inflammatory bowel disease. AML patients with neutropenic colitis suffer from a condition which is pathophysiologically closely related to the studied diseases. It is therefore reasonable to raise the question whether this cohort would equally benefit from a novel nutritional regimen enriched in omega-3 PUFA.

The proposed pilot study will address the question of the clinical value of adding an omega-3 PUFA containing lipid emulsion to the TPN regimen as regards protection against colitis ≥ °3 (primary objective). A numerical cutoff will be provided to support the decision whether further investigation is warranted or the intervention is considered not promising.

Target accrual is n=35 patients receiving TPN. An interim analysis will be performed after n1=13 patients will be evaluable for the primary endpoint. The results of this interim analysis will determine whether continuation of the trial is of interest or the trial be stopped. The sample size has been calculated by the use of Simon's two-stage minimax design.

ELIGIBILITY:
Inclusion Criteria:

* All of the following:

Subjects with a cyto- or histopathologically confirmed diagnosis of newly diagnosed:

* AML or
* biphenotypic acute leukemia with predominantly myeloid features undergoing myeloablative treatment analogous to AML or
* refractory anemia with excess of blasts (RAEB) or refractory anemia with excess of blasts in transformation (RAEB-t) with an IPSS score of >1.5 (appendix 10.8.) and

  * ECOG performance status (PS) £2 (see appendix 10.2.) and
  * Written informed consent

Exclusion Criteria:

One or more of the following:

* Contraindication to myeloablative chemotherapy, intravenous lipids, or TPN
* Previous or concomitant chronic inflammatory bowel disease, unspecified colitis or pancreatitis
* Impaired hepatic or renal function as defined by:

  * ALAT and/or ASAT >3 x upper normal limit (UNL) and/or Bilirubin >3 x UNL unless increase is most likely caused by AML organ infiltration
  * Serum creatinin >3 x UNL (after adequate hydration), unless increase is most likely caused by AML organ infiltration
* Other concurrent severe and/or uncontrolled medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
efficacy of an omega-3 PUFA containing lipid emulsion in reducing the incidence of °3-4 colitis (CTC AE v3.0) | time to completion of cytotoxic chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Bükki, MD, Principal Investigator — Inselspital Berne
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Bukki J, Stanga Z, Tellez FB, Duclos K, Kolev M, Krahenmann P, Pabst T, Iff S, Juni P. Omega-3 poly-unsaturated fatty acids for the prevention of severe neutropenic enterocolitis in patients with acute myeloid leukemia. Nutr Cancer. 2013;65(6):834-42. doi: 10.1080/01635581.2013.801998. PMID 23909727